CLINICAL TRIAL: NCT05801003
Title: Cutting Balloon Predilation Prior to Abluminus Sirolimus-eluting Stent Implantation
Brief Title: Cutting Balloon Predilation Prior to Abluminus Sirolimus-eluting Stent Implantation (CUT-DRESS).
Acronym: CUT-DRESS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario La Fe (Other)
Responsible Party: Principal Investigator, Jorge Sanz Sanchez, Specialist in Cardiology, MD, PhD, Hospital Universitario La Fe
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 529
Record Dates: First submitted 2023-03-11; First posted 2023-04-06 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Coronary Artery Disease; Percutaneous Coronary Intervention; Cutting Balloon
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, randomized controlled trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Pre-dilation with cutting balloon followed by ASES implantation.
  Interventions: Device: Predilation with cutting balloon.
- Control group (Active Comparator): Pre-dilation with a standard balloon (semi-compliant or non-compliant) followed by ASES implantation.
  Interventions: Device: Predilation with conventional balloon

INTERVENTIONS:
Device: Predilation with cutting balloon. — PCI will be performed under OCT guidance. Predilation of the lesion will be done with cutting balloon.
  Other Names: Wolverine Cutting balloon
  Arms: Study group
Device: Predilation with conventional balloon — PCI will be performed under OCT guidance. Predilation of the lesion will be done with conventional balloon (semi-compliant or non-compliant)
  Arms: Control group

SUMMARY:
Drug-eluting stents iterations has significantly improved the results of percutaneous revascularization among patients undergoing coronary revascularization thanks to thinner struts, more biocompatible polymer coatings and new drug release formulations; leading to lower thrombogenicity, faster reendothelialization and improved clinical outcomes. Notwithstanding, stent-related events yet occur.

Lesion pre-dilation prior to DES implantation is a crucial procedural step as it creates microdissections, which are required for optimal uptake of the drug. However, the best pre-dilation strategy has not yet been determined. Therefore, the aim of this study is to evaluate a strategy based on pre-dilation with cutting balloon (CB) followed by Abluminus Sirolimus-eluting stent (ASES) implantation for de novo coronary lesions

DETAILED DESCRIPTION:
The study will be a prospective, multicenter, randomized controlled trial in patients undergoing PCI with the novo coronary disease.

A total of 96 patients with de novo coronary artery stenosis will be included.

After being informed about the study and the potential risks, all patients meeting all the inclusion criteria and none of exclusion criteria will give written informed consent. Random allocation in a 1:1 fashion to one of the following strategies:

A) Study group: Pre-dilation with cutting balloon followed by ASES implantation.

B) Control group: Pre-dilation with a standard balloon (semi-compliant or non-compliant) followed by ASES implantation.

Stent optimisation will be performed based on intracoronary imaging findings.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic coronary artery disease or evidence of ischemia in the presence of one or more coronary artery stenoses >50% in a native coronary artery.

Exclusion Criteria:

1. Cardiogenic shock
2. Patients presenting with ST-segment elevation myocardial infarction
3. Patients undergoing chronic total occlusions PCI
4. Patients undergoing left main PCI
5. Patients undergoing venous bypass graft lesions PCI
6. Patients with in-stent restenosis
7. Inability to provide informed consent
8. Life expectancy <1year due to non-cardiac disease
9. Currently participating in another trial before reaching first endpoint

There will be no exclusion based on mode of co-morbidities, left ventricular function, number of diseased vessels and lesions, or number of target lesions.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Minimum stent area post-stenting measured by optimal coherence tomography (OCT) | Immediately after the procedure

SECONDARY OUTCOMES:
Percentage of neointimal hyperplasia (%) measured by OCT coherence tomography (OCT). | 9 month follow-up.
  Key secondary
Mean stent area measured by optimal coherence tomography | 9 month follow-up.
Acute procedural success | Immediately after the procedure
Coronary disection | Immediately after the procedure
Malapposition (Major/minor) post-stenting measured by optimal coherence tomography | Immediately after the procedure and at 9 month follow-up
Mean neointimal hyperplasia area measured by optimal coherence tomography | 9 months
Minimum stent eccentricity measured by optimal coherence tomography | 9 months
Stent asymmetry index measured by optimal coherence tomography | 9 months
All cause death | 12 months
Death from cardiovascular causes | 12 months
Target vessel myocardial infarction | 12 months
Target lesion revascularization | 12 months
Stent thrombosis | 12 months
Any myocardial infarction | 12 months

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario y Politécnico La Fe, Valencia
  - Hospital General de Valencia, Valencia